CLINICAL TRIAL: NCT03704831
Title: Comparison of Analgesic Efficiency Between IPACK Block (Interspace Between the Popliteal Artery and the Capsule of the Posterior Knee) and Surgical Infiltration After Total Knee Arthroplasty
Brief Title: Comparison of Analgesic Efficiency Between IPACK Block and Surgical Infiltration After Total Knee Arthroplasty
Acronym: IPACK
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL18_0304
Record Dates: First submitted 2018-09-24; First posted 2018-10-15 (Actual); Last update posted 2020-03-10 (Actual); Status verified 2020-03

CONDITIONS: Total Knee Arthroplasty
Keywords: Locoregional anesthesia; IPACK block; surgical infiltration; Total knee arthroplasty

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- IPACK group: IPACK group
  Interventions: Other: Injection of local anesthetics during total knee arthroplasty by a locoregional anesthesia named IPACK block
- Surgical infiltration group: Surgical infiltration group
  Interventions: Other: Injection of local anesthetics during total knee arthroplasty by surgical infiltration

INTERVENTIONS:
Other: Injection of local anesthetics during total knee arthroplasty by a locoregional anesthesia named IPACK block — Injection of local anesthetics during total knee arthroplasty by a locoregional anesthesia named IPACK block (Interspace between the Popliteal Artery and the Capsule of the posterior Knee)
  Groups: IPACK group
Other: Injection of local anesthetics during total knee arthroplasty by surgical infiltration — Injection of local anesthetics during total knee arthroplasty by surgical infiltration.
  Groups: Surgical infiltration group

SUMMARY:
The purpose of this retrospective study is to compare the analgesic efficiency of IPACK block (Interspace between the Popliteal Artery and the Capsule of the posterior Knee) with surgical infiltration after total knee arthroplasty. The main objective is to compare cumulative morphine consumption the first 24 hours after surgery. The secondary objectives are to compare pain scores, types and amounts of other analgesics needed during the first 24 hours after surgery.

DETAILED DESCRIPTION:
After patient agreement, data will be collected on patient records and will be compared into 2 groups.

Data will be :

* cumulative consumption of morphine during the first 24 hours after surgery
* pain scores during the first 24 hours after surgery
* amount of analgesics during the first 24 hours after surgery
* maximal pain score during the first 24 hours after surgery

ELIGIBILITY:
Inclusion criteria:

- All adults patients after a total knee arthroplasty since november 2015

Exclusion criteria:

- Child, non primitive surgery

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All adults patients after a total knee arthroplasty
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2018-10-20 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2019-11-30 (Actual)

PRIMARY OUTCOMES:
Analgesic need | 24 hours
  Morphine consumption during the first 24 hours after total knee arthroplasty

SECONDARY OUTCOMES:
Pain scores in the recovery room | 24 hours
  Pain scores in the recovery room during the first 24 hours after surgery using the EVA scale
maximal pain score | 24 hours
  maximal pain score during the first 24 hours after surgery using the EVA scale
Description of the analgesics administered | 24 hours
  types of other analgesics needed during the first 24 hours after surgery
amount other analgesics | 24 hours
  amount other analgesics needed during the first 24 hours after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Xavier Capdevila, PhD, Study Director — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France